CLINICAL TRIAL: NCT02958241
Title: Supine vs. Upright Weight Bearing MRI in the Evaluation of Patients With Lumbar Spondylolisthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Texas Back Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRI001
Record Dates: First submitted 2016-11-03; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Spondylolisthesis
Keywords: spondylolisthesis; Lumbar spine; MRI
MeSH Terms: conditions — Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MRI — Supine and weight bearing MRI

SUMMARY:
This study investigates the possible differences in images obtained in patients with lumbar spondylolisthesis when positioned in an upright weight bearing position compared with traditional supine positioning for lumbar MRI.

DETAILED DESCRIPTION:
Detailed Description Spondylolisthesis is a spinal condition in which one vertebral body has slid forward in relation to the vertebrae below and is sometimes associated with spinal instability. Lumbar spondylolisthesis is a relatively common problem and is generally diagnosed from radiographs. MRI is often used to evaluate the condition further and to determine if there is nerve root compression involved. One potential disadvantage with traditional MRI to evaluate spondylolisthesis is imaging is performed with the patient lying supine in the scanner. This creates a potential for the superior vertebra to slide posteriorly so that the extent of the slip may not be fully appreciated, if seen at all. Use of upright weight bearing MRI provides the opportunity to image the spine in the position that patients are most likely to experience symptoms and is similar to standing radiographs.

MRI Acquisition: Each patient will undergo MRI scanning in the supine and weight bearing positions during the same imaging session. If it is determined that a patient who has consented to participate in the study should not have an MRI made due to safety concerns (such as metallic implant or other contraindication to MRI not identified during recruiting), they will be discontinued from the study and another patient recruited to fulfill the planned number of images available for analysis.

The MRI procedure will be standard lumbar spine scanning protocol using the Esaote G-scan, an open unit. Patients will be scanned supine and then the unit rotated to 81 degrees from horizontal for the weight bearing scan. Immediately after each scan, the patient will complete visual analog scales (VAS) assessing back and leg pain.

Researcher(s) performing image assessments will be blinded to the position in which scans were made. Data to be recorded for each image is the Meyerding scale (1-4 scale rating the severity of the spondylolisthesis), amount of slip (mm), anterior and posterior disc space height (mm), foraminal area, anteroposterior (AP) distance at the most narrow part of the foramen, and disc space angulation. Area of the spinal canal and AP distance across the canal will be measured from axial images. The facet fluid sign, associated with spinal instability, will be assessed from axial MRI views using a 3-point scale with "none" indicating no evidence of fluid in the left or right facet joints; "possible" if there is some suggestion of fluid in the joints; or "definite" if there is at least a 2 mm wide layer of hyperintensity within either joint bilaterally at the level evaluated. Additionally, the width of the fluid fill of the facet joint taken perpendicular to the apparent joint line, and the largest value recorded as effusion size.

Clinical Assessments: VAS separately assessing back and leg pain will be completed immediately after the supine scanning and again immediately after weight bearing scanning. Analysis will be conducted to determine if differences in pain correlate with changes in images taken in the two positions.

Statistical methods: Parametric measures will be compared for the two imaging positions using paired t-tests. Pairwise categorical data will be analyzed using McNemar analysis. In the secondary study dealing with facet fluid sign, mean values for translation, disc height, foraminal area, and AP distance will be compared across the three facet fluid sign categories using ANOVA.

Changes in back and leg pain will be analyzed to determine if there is a relationship between these changes and changes noted on the positional MRI. It is not anticipated that this section of the study will produce statistically significant results, but will hopefully provide guidance for possibly investigating these parameters in future studies.

From routine clinical lateral flexion/extension radiographs, change in translation between the two positions will be measured. If a lateral neutral radiograph is available, translation as well as anterior and posterior disc height will be measured. All measurements will be made using the same methods as described for the MRIs.

Sample size: At least 25 patients, but no more than 60 patients will be included. After 25 patients are imaged, data will be analyzed to determine an appropriate sample size to determine a statistically significant difference between measurements made from the supine and upright weight bearing images.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of degenerative or isthmic lumbar spondylolisthesis by a spine specialty physician based on clinical evaluation and lumbar radiographs
* No previous lumbar spinal fusion at the level of the spondylolisthesis or a procedure resulting in the presence of metallic implants at the level of interest (if a device such as a interspinous device was implanted and later removed, the patient may participate in the study)
* Be able and willing to provide written consent to participate in the study
* Willing to undergo a second MRI approximately 6 months after surgery, if surgery is performed

Exclusion Criteria:

* Pregnancy
* Any condition that would prevent the patient from undergoing MRI
* Recent lumbar vertebral body fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Superior vertebral body translation (mm) | up to 6 months
Disc space height (mm) | up to 6 months

SECONDARY OUTCOMES:
Foraminal area (mm2) | initial evaluation and 6 mo after surgery if surgery is performed
Meyerding grade and facet fluid fill sign (value assigned based on visual inspecting of the MRIs and applying published scoring grades) | initial evaluation and 6 mo after surgery if surgery is performed
Visual analog pain scales (VAS) assessing back and leg pain | initial evaluation and 6 mo after surgery if surgery is performed
Anteroposterior distance across spinal canal (mm) | initial evaluation and 6 mo after surgery if surgery is performed
Spinal canal area (mm2) | initial evaluation and 6 mo after surgery if surgery is performed

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Back Institute, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No